CLINICAL TRIAL: NCT01972529
Title: A Randomized, Global, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Once-daily Oral Avatrombopag for the Treatment of Adults With Thrombocytopenia Associated With Liver Disease Prior to an Elective Procedure
Brief Title: Treatment of Thrombocytopenia in Patients With Chronic Liver DiseaseUndergoing an Elective Procedure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E5501-G000-310; 2013-000965-34 (EudraCT Number)
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Results first posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-01

CONDITIONS: Thrombocytopenia Associated With Liver Disease
Keywords: Thrombocytopenia; Chronic Liver Disease
MeSH Terms: conditions — Thrombocytopenia | interventions — avatrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (avatrombopag, lower baseline platelet count) (Experimental): 60 mg avatrombopag (3 x 20 mg tablets) once daily on Days 1 through 5
  Interventions: Drug: avatrombopag (lower baseline platelet count)
- Group B (placebo, lower baseline platelet count) (Placebo Comparator): placebo (3 x 20 mg matching placebo tablets) once daily on Days 1 through 5
  Interventions: Drug: placebo (lower baseline platelet count)
- Group C (avatrombopag, higher baseline platelet count) (Experimental): 40 mg avatrombopag (2 x 20 mg tablets) once daily on Days 1 through 5
  Interventions: Drug: avatrombopag (higher baseline platelet count)
- Group D (placebo, higher baseline platelet count) (Placebo Comparator): placebo (2 x 20 mg matching placebo tablets) once daily on Days 1 through 5
  Interventions: Drug: placebo (higher baseline platelet count)

INTERVENTIONS:
Drug: avatrombopag (lower baseline platelet count) — 60 mg avatrombopag (3 x 20 mg tablets)
  Arms: Group A (avatrombopag, lower baseline platelet count)
Drug: placebo (lower baseline platelet count) — 60 mg placebo (3 x 20 mg matching placebo tablets)
  Arms: Group B (placebo, lower baseline platelet count)
Drug: avatrombopag (higher baseline platelet count) — 40 mg avatrombopag (2 x 20 mg tablets)
  Arms: Group C (avatrombopag, higher baseline platelet count)
Drug: placebo (higher baseline platelet count) — 40 mg placebo (2 x 20 mg matching placebo tablets)
  Arms: Group D (placebo, higher baseline platelet count)

SUMMARY:
This is a global, multicenter, randomized, double-blind, placebo-controlled, parallel group study using avatrombopag to treat adults with thrombocytopenia associated with liver disease. The study will evaluate avatrombopag in the treatment of thrombocytopenia associated with liver disease prior to an elective procedure to reduce the need for platelet transfusions or any rescue procedure for bleeding due to procedural and post-procedural bleeding complications. Participants will be enrolled into 2 cohorts according to mean baseline platelet count and, within each baseline platelet count cohort will be further stratified by risk of bleeding associated with the elective procedure (low, moderate, or high) and hepatocellular carcinoma (HCC) status (Yes or No).

DETAILED DESCRIPTION:
This study will consist of 3 phases: Prerandomization, Randomization, and a Follow-up Phase. The Prerandomization Phase includes one Screening Visit that will take place from Day -14 through Day -1; the Randomization Phase includes the Baseline Period, Treatment Period, and Procedure Day Period (5 to 8 days after last dose of study drug [Study Day 10 to 13]). The Follow-up Phase comprises 2 visits: 7 days post Procedure Day and 30 days after receiving the last dose of study drug. Permitted procedures include: Paracentesis; Thoracentesis; Gastrointestinal endoscopy with or without plans for biopsy, colonoscopy, polypectomy, or variceal banding; Liver biopsy; Bronchoscopy with or without plans for biopsy; Ethanol ablation therapy or chemoembolization for HCC; Vascular catheterization (including right side procedures in participants with pulmonary hypertension); Transjugular intrahepatic portosystemic shunt; Dental procedures; Renal biopsy; Biliary interventions; Nephrostomy tube placement; Radiofrequency ablation; and Laparoscopic interventions.

ELIGIBILITY:
Inclusion Criteria

1. Participants greater than or equal to 18 years of age at Screening with chronic liver disease
2. Participants who have a mean baseline platelet count of less than 50 x 10^9/L. Platelet counts must be measured on 2 separate occasions, during the Screening Period and at Baseline, and must be performed at least one day apart with neither platelet count greater than 60 x 10^9/L. The mean of these 2 platelet counts (mean baseline platelet count) will be used for entry criteria and for assignment to the low or high baseline platelet count cohort.
3. Participants scheduled to undergo a permitted elective procedure who, in the opinion of the investigator, will require a platelet transfusion to address a risk of bleeding associated with the procedure unless there is a clinically significant increase in platelet count from baseline
4. Model For End-stage Liver Disease (MELD) score less than or equal to 24 at Screening
5. If taking inhibitors of P glycoprotein (P-gp), except for verapamil, dose must be stable for 7 days prior to Screening
6. Provide written informed consent
7. Willing and able to comply with all aspects of the protocol

Exclusion Criteria

1. Any history of arterial or venous thrombosis, including partial or complete thrombosis
2. Evidence of thrombosis (partial or complete) in the main portal vein, portal vein branches, or any part of the splenic mesenteric system at Screening
3. Portal vein blood flow velocity rate <10 centimeters/second at Screening
4. Hepatic encephalopathy that cannot be effectively treated
5. Participants with HCC with Barcelona Clinic Liver Cancer (BCLC) staging classification C or D
6. Platelet transfusion or receipt of blood products containing platelets within 7 days of Screening. However packed red blood cells are permitted.
7. Heparin, warfarin, nonsteroidal anti-inflammatory drugs (NSAID), aspirin, verapamil, and antiplatelet therapy with ticlopidine or glycoprotein IIb/IIIa antagonists (eg, tirofiban) within 7 days of Screening
8. Use of erythropoietin stimulating agents within 7 days of Screening
9. Interferon (IFN) use within 14 days of Screening
10. Estrogen-containing hormonal contraceptive or hormone replacement therapy use within 30 days of Screening
11. Active infection requiring systemic antibiotic therapy within 7 days of Screening. However, prophylactic use of antibiotics is permitted.
12. Alcohol abuse, alcohol dependence syndrome, drug abuse, or drug dependence within 6 months of the study start (unless participating in a controlled rehabilitation program) or acute alcoholic hepatitis (chronic alcoholic hepatitis is allowed) within 6 months of the study start
13. Elective procedure performed prior to Visit 4 (Procedure Day)
14. Known to be human immunodeficiency virus positive
15. Any clinically significant acute or active bleeding (eg, gastrointestinal, central nervous system)
16. Known history of any primary hematologic disorder (eg, immune thrombocytopenic purpura, myelodysplastic syndrome)
17. Known medical history of genetic prothrombotic syndromes (eg, Factor V Leiden; prothrombin G20210A; ATIII deficiency, etc.)
18. Participants with a history of significant cardiovascular disease (eg, congestive heart failure New York Heart Association Grade III/IV, arrhythmia known to increase the risk of thromboembolic events [eg, atrial fibrillation], coronary artery stent placement, angioplasty, and coronary artery bypass grafting)
19. Females of childbearing potential who have had unprotected sexual intercourse within 30 days before study entry and who do not agree to use a highly effective method of contraception (eg, total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a progesterone-only contraceptive implant/injection, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation. If currently abstinent, the participant must agree to use a double-barrier method as described above if she becomes sexually active during the study period or for 30 days after study drug discontinuation. All females will be considered to be of childbearing potential unless they are postmenopausal (at least 12 months consecutive amenorrhea in the appropriate age group and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, hysterectomy, or bilateral oophorectomy) at least 1 month before dosing.
20. Females who are lactating or pregnant at Screening or Baseline (as documented by a positive serum beta-human chorionic gonadotropin [B-hCG] test with a minimum sensitivity 25 IU/L or equivalent units of B-hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
21. Post liver transplant participants
22. Any participant who has previously received avatrombopag
23. Hypersensitivity to avatrombopag maleate or any of its excipients
24. Hemoglobin levels ≤ 8.0 or ≥ 18.0 g/dL for men and > 15 for women at Screening, with hematocrit ≥ 54% for men and ≥ 45% for women
25. Current malignancy including solid tumors and hematologic malignancies (except HCC)
26. Any history of concomitant medical condition that, in the opinion of the investigator(s), would compromise the participant's ability to safely complete the study
27. Currently enrolled in another clinical trial with any investigational drug or device within 30 days of Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-01-26 (Actual); Study Completion 2017-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (109):
- United States (21):
  - Lancaster, California
  - Long Beach, California
  - Los Angeles, California
  - Sacramento, California
  - San Bernardino, California
  - San Francisco, California
  - Jacksonville, Florida
  - Palmetto Bay, Florida
  - Tampa, Florida
  - New Orleans, Louisiana
  - Rochester, Michigan
  - Minneapolis, Minnesota
  - Jackson, Mississippi
  - New York, New York
  - The Bronx, New York
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
  - Harlingen, Texas
  - Houston, Texas
  - San Antonio, Texas
- Argentina (3):
  - Pilar, Buenos Aires
  - Ciudad Autonoma Buenos Aires
  - Mendoza
- Australia (3):
  - Camperdown, New South Wales
  - Adelaide, South Australia
  - Bedford Park, South Australia
- Austria (2):
  - Linz
  - Vienna
- Belgium (2):
  - Brussels
  - Leuven
- Brazil (3):
  - Porto Alegre, Rio Grande do Sul
  - São José do Rio Preto, São Paulo
  - São Paulo
- Canada (2):
  - London, Ontario
  - Toronto, Ontario
- Chile (2):
  - La Serena
  - Santiago
- China (4):
  - Changsha, Hu'nan
  - Nanjing, Jiangsu
  - Shanghai, Shanghai Municipality
  - Beijing
- France (6):
  - Strasbourg, Bas Rhin
  - Grenoble, Isere
  - Reims, Marne
  - Clermont-Ferrand, Puy De Dome
  - Amiens, Somme
  - Vandœuvre-lès-Nancy
- Germany (5):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Cologne, North Rhine-Westphalia
  - Herne, North Rhine-Westphalia
  - Kiel, Schleswig-Holstein
  - Hamburg
- Hungary (8):
  - Békéscsaba
  - Budapest
  - Dunaújváros
  - Gyula
  - Kaposvár
  - Kecskemét
  - Szombathely
  - Zalaegerszeg
- Italy (8):
  - San Giovanni Rotondo, Foggia
  - Bari
  - Bologna
  - Genova
  - Milan
  - Modena
  - Palermo
  - Udine
- Poland (5):
  - Katowice
  - Lodz
  - Mysłowice
  - Szczecin
  - Wroclaw
- Portugal (6):
  - Coimbra
  - Lisbon
  - Porto
  - Viana do Castelo
  - Vila Real
  - Viseu
- South Korea (10):
  - Chuncheon, Gangwon-do
  - Guri-si, Gyeonggi-do
  - Seongnam-si, Gyeonggi-do
  - Suwon, Gyeonggi-do
  - Yangsan, Gyeongsangnam-do
  - Hwasun, Jeollanam-do
  - Busan
  - Daegu
  - Incheon
  - Seoul
- Spain (5):
  - Barcelona
  - Pontevedra
  - Seville
  - Valencia
  - Valladolid
- Taiwan (5):
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan
- Thailand (4):
  - Bangkoknoi, Bangkok
  - Ratchathewi, Bangkok
  - Khlong Luang, Changwat Pathum Thani
  - Mueang Nonthaburi, Chiang Mai
- United Kingdom (5):
  - Truro, Cornwall
  - London, Greater London
  - Manchester, Greater Manchester
  - Wolverhampton, West Midlands
  - Leeds, West Yorkshire

REFERENCES:
- [Derived] Poordad F, Terrault NA, Alkhouri N, Tian W, Allen LF, Rabinovitz M. Avatrombopag, an Alternate Treatment Option to Reduce Platelet Transfusions in Patients with Thrombocytopenia and Chronic Liver Disease-Integrated Analyses of 2 Phase 3 Studies. Int J Hepatol. 2020 Jan 25;2020:5421632. doi: 10.1155/2020/5421632. eCollection 2020. PMID 32047671
- [Derived] Terrault N, Chen YC, Izumi N, Kayali Z, Mitrut P, Tak WY, Allen LF, Hassanein T. Avatrombopag Before Procedures Reduces Need for Platelet Transfusion in Patients With Chronic Liver Disease and Thrombocytopenia. Gastroenterology. 2018 Sep;155(3):705-718. doi: 10.1053/j.gastro.2018.05.025. Epub 2018 May 17. PMID 29778606

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 370 participants signed informed consent. Of these 370 participants, 139 were screening failures and 231 were randomized into the study. Of the 139 screening failures, 120 did not meet the inclusion/exclusion criteria and the other 19 participants failed due to adverse events, lost to follow-up and withdrawal of consent.
Groups:
- 60 mg Placebo (Lower Baseline Platelet Count): Participants with a baseline platelet count of less than 40 x 10^9/liters (L) took three 20 milligrams (mg) (60 mg total) matching placebo tablets orally, once daily with a meal during the Treatment Period on Days 1 through 5, and 5 to 8 days prior to the scheduled procedure.
- 60 mg Avatrombopag, (Lower Baseline Platelet Count): Participants with a baseline platelet count of less than 40 x 10^9/L took three 20 mg tablets (60 mg total) avatrombopag (2nd generation) orally, once daily with a meal during the Treatment Period on Days 1 through 5, and 5 to 8 days prior to the elective procedure.
- 40 mg Placebo (Higher Baseline Platelet Count): Participants with a baseline platelet count of greater than or equal to 40 to less than 50 x 10^9/L took two 20 mg matching placebo tablets orally, once daily with a meal during the Treatment Period on Days 1 through 5, and 5 to 8 days prior to the scheduled procedure.
- 40 mg Avatrombopag (Higher Baseline Platelet Count): Participants with a baseline platelet count of greater than or equal to 40 to less than 50 x 10^9/L took two 20 mg tablets (40 mg total) avatrombopag (2nd generation) orally, once daily with a meal during the Treatment Period on Days 1 through 5, and 5 to 8 days prior to the scheduled procedure.
Period: Overall Study
Arm/Group | 60 mg Placebo (Lower Baseline Platelet Count) | 60 mg Avatrombopag, (Lower Baseline Platelet Count) | 40 mg Placebo (Higher Baseline Platelet Count) | 40 mg Avatrombopag (Higher Baseline Platelet Count)
Started | 48 | 90 | 34 | 59
Completed | 46 | 85 | 32 | 55
Not Completed | 2 | 5 | 2 | 4
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Participant Choice | 0 | 1 | 0 | 0
Not completed — Withdrawl of Consent | 1 | 2 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 2
Not completed — Not treated | 0 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set was defined as the group of all randomized participants.
Groups:
- 60 mg Placebo (Lower Baseline Platelet Count): Participants with a baseline platelet count of less than 40 x 10^9/liters (L) took three 20 milligrams (mg) matching placebo tablets orally, once daily with a meal during the Treatment Period on Days 1 through 5, and 5 to 8 days prior to the scheduled procedure.
- 60 mg Avatrombopag, (Lower Baseline Platelet Count): Participants with a baseline platelet count of less than 40 x 10^9/L took three 20 mg tablets (60 mg total) avatrombopag (2nd generation) orally, once daily with a meal during the Treatment Period on Days 1 through 5, and 5 to 8 days prior to the scheduled procedure.
- Total: Total of all reporting groups
Arm/Group | 60 mg Placebo (Lower Baseline Platelet Count) | 60 mg Avatrombopag, (Lower Baseline Platelet Count) | 40 mg Placebo (Higher Baseline Platelet Count) | 40 mg Avatrombopag (Higher Baseline Platelet Count) | Total
Number analyzed (Participants) | 48 | 90 | 34 | 59 | 231
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.1 (11.02) | 55.6 (9.12) | 57.8 (11.05) | 57.5 (10.06) | 56.3 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 25 | 10 | 22 | 73
  Male | 32 | 65 | 24 | 37 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 3 | 7 | 30
  Not Hispanic or Latino | 37 | 77 | 31 | 51 | 196
  Unknown or Not Reported | 1 | 3 | 0 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 18 | 32 | 15 | 24 | 89
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 0 | 2 | 5
  White | 28 | 50 | 19 | 31 | 128
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 0 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Did Not Require a Platelet Transfusion or Any Rescue Procedure for Bleeding After Randomization Following a Scheduled Procedure
Description: Responders were defined as participants who did not require a platelet transfusion or any rescue procedure for bleeding after randomization and up to 7 days following a scheduled procedure. Participants with missing information due to early withdrawal or other reasons were conservatively considered as having received a transfusion in the analysis, (i.e. a Non-responder).
Time Frame: Baseline (Visit 2) up to 7 days following a scheduled procedure
Population: Full analysis Set (FAS) was defined as the group of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- 60 mg Placebo (Lower Baseline Platelet Count): Participants with a baseline platelet count of less than 40 x 10^9/liters (L ) took three 20 milligrams (mg) matching placebo tablets orally, once daily with a meal during the Treatment Period on Days 1 through 5, and 5 to 8 days prior to the scheduled procedure.
Arm/Group | 60 mg Placebo (Lower Baseline Platelet Count) | 60 mg Avatrombopag, (Lower Baseline Platelet Count) | 40 mg Placebo (Higher Baseline Platelet Count) | 40 mg Avatrombopag (Higher Baseline Platelet Count)
Number analyzed (Participants) | 48 | 90 | 34 | 59
Percentage of participants | 22.9 [11.0 to 34.8] | 65.6 [55.7 to 75.4] | 38.2 [21.9 to 54.6] | 88.1 [79.9 to 96.4]
Statistical Analysis 1: Comparison: 60 mg Placebo (Lower Baseline Platelet Count) vs 60 mg Avatrombopag, (Lower Baseline Platelet Count); The null hypothesis was that the proportion of participants not requiring a platelet transfusion or any rescue procedure for bleeding after randomization and up to 7 days following a scheduled procedure was the same between the 60 mg avatrombopag and matched placebo treatment groups; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by the risk of bleeding associated with the elective procedure within each baseline platelet count cohort; Difference of proportion vs placebo = 42.6, 95% CI 2-sided [27.2 to 58.1] — Difference of proportion versus (vs) placebo = proportion of Responders for avatrombopag - proportion of Responders for placebo; 95% CI is calculated based on normal approximation
Statistical Analysis 2: Comparison: 40 mg Placebo (Higher Baseline Platelet Count) vs 40 mg Avatrombopag (Higher Baseline Platelet Count); The null hypothesis was that the proportion of participants not requiring a platelet transfusion or any rescue procedure for bleeding after randomization and up to 7 days following a scheduled procedure was the same between the avatrombopag and placebo treatment groups; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by the risk of bleeding associated with the elective procedure within each baseline platelet count cohort; Difference of proportion vs placebo = 49.9, 95% CI 2-sided [31.6 to 68.2] — Difference of proportion vs placebo = proportion of Responders for avatrombopag - proportion of Responders for placebo; 95% CI is calculated based on normal approximation

2. Secondary Outcome: Percentage of Participants Who Achieved a Platelet Count Greater Than or Equal to 50 x 10^9/L on the Scheduled Procedure Day
Description: Responders were defined as participants who achieved a platelet count greater than or equal to 50 x 10^9/L on the procedure day. Participants with missing a platelet count on the procedure day were conservatively considered as not achieving a platelet count of 50x10^9/L in the analysis, (i.e. Non-responders).
Time Frame: Day 10 to Day 13 (Visit 4)
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- 60 mg Placebo (Lower Baseline Platelet Count): Participants with a baseline platelet count of less than 40 x 10^9/L took three 20 mg matching placebo tablets orally, once daily with a meal during the Treatment Period on Days 1 through 5, and 5 to 8 days prior to the scheduled procedure.
Arm/Group | 60 mg Placebo (Lower Baseline Platelet Count) | 60 mg Avatrombopag, (Lower Baseline Platelet Count) | 40 mg Placebo (Higher Baseline Platelet Count) | 40 mg Avatrombopag (Higher Baseline Platelet Count)
Number analyzed (Participants) | 48 | 90 | 34 | 59
Percentage of participants | 4.2 [0.0 to 9.8] | 68.9 [59.3 to 78.5] | 20.6 [7.0 to 34.2] | 88.1 [79.9 to 96.4]
Statistical Analysis 1: Comparison: 60 mg Placebo (Lower Baseline Platelet Count) vs 60 mg Avatrombopag, (Lower Baseline Platelet Count); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; P-value is stratified by the risk of bleeding associated with the elective procedure within each baseline platelet count cohort; Difference of proportion vs placebo = 64.7, 95% CI 2-sided [53.6 to 75.8] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: 40 mg Placebo (Higher Baseline Platelet Count) vs 40 mg Avatrombopag (Higher Baseline Platelet Count); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Difference of percentage vs placebo = 67.5, 95% CI 2-sided [51.6 to 83.4] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Change From Baseline in Platelet Count on the Scheduled Procedure Day
Description: Last observation carried forward was used for participants with a missing platelet count on the scheduled procedure day. Platelet count was measured preprocedure and before any platelet transfusion.
Time Frame: Baseline (Visit 2) to Procedure Day 10 to Day 13 (Visit 4)
Population: FAS
Measure: Mean (Standard Deviation); unit: Platelet count x 10^9/per liter
Arm/Group | 60 mg Placebo (Lower Baseline Platelet Count) | 60 mg Avatrombopag, (Lower Baseline Platelet Count) | 40 mg Placebo (Higher Baseline Platelet Count) | 40 mg Avatrombopag (Higher Baseline Platelet Count)
Number analyzed (Participants) | 48 | 88 | 32 | 58
Platelet count x 10^9/per liter | 0.8 (6.36) | 32.0 (25.53) | 1.0 (9.30) | 37.1 (27.41)
Statistical Analysis 1: Comparison: 60 mg Placebo (Lower Baseline Platelet Count) vs 60 mg Avatrombopag, (Lower Baseline Platelet Count); Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney); P-value is based on Wilcoxon rank sum test for each avatrombopag treatment group vs placebo within each baseline platelet count cohort; Difference in change of platelet count = 27.5, 95% CI 2-sided [22.5 to 32.5] — Difference in change from baseline of platelet count for avatrombopag vs placebo within each baseline platelet count cohort is based on Hodges-Lehmann estimation; 95% confidence interval is the asymptotic (Moses) CI
Statistical Analysis 2: Comparison: 40 mg Placebo (Higher Baseline Platelet Count) vs 40 mg Avatrombopag (Higher Baseline Platelet Count); Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney); [statistical method as in outcome 3, analysis 1]; Difference in change of platelet count = 33.0, 95% CI 2-sided [25.5 to 41.5] — [estimate comment as in outcome 3, analysis 1]

4. Other Pre Specified Outcome: Percentage of Participants With a World Health Organization (WHO) Bleeding Score Greater Than or Equal to 2 After a Scheduled Procedure
Description: The severity of bleeding events was assessed by the investigator (or appropriately delegated study site personnel) using the WHO bleeding scale. The WHO bleeding scale is a clinical investigator-assessed five-point scale with Grade 0 = No bleeding, Grade 1 = Petechial bleeding, Grade 2 = Mild blood loss (clinically significant), Grade 3 = Gross blood loss (requires transfusion (severe)), and Grade 4 = Debilitating blood loss, retinal or cerebral associated with fatality. Participants with missing information are considered as having a WHO bleeding score greater than or equal to 2 in the analysis.
Time Frame: Baseline (Visit 2) up to 7 days post scheduled procedure
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | 60 mg Placebo (Lower Baseline Platelet Count) | 60 mg Avatrombopag, (Lower Baseline Platelet Count) | 40 mg Placebo (Higher Baseline Platelet Count) | 40 mg Avatrombopag (Higher Baseline Platelet Count)
Number analyzed (Participants) | 48 | 90 | 34 | 59
Percentage of participants | 6.3 | 5.6 | 2.9 | 0

5. Other Pre Specified Outcome: Number of Participants Experiencing an Adverse Event
Description: Safety assessments consisted of monitoring and recording all adverse events (AEs) and serious adverse events, including platelet transfusion-related complications; routine laboratory evaluation for hematology, serum chemistry, and urine values; periodic measurement of vital signs and electrocardiograms (ECGs); the performance of physical examinations; and Doppler sonography. AE severity was graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, where Grade 1 = mild, Grade 2 = moderate, Grade 3 = Severe, Grade 4 = Life-threatening, and Grade 5 = Death related to the AE. All AEs graded as 4 or 5 were considered to be serious. Treatment-emergent adverse events (TEAEs) were defined as an AE that started on or after the date of first dose of study drug, up to 30 days after the last dose of study drug. Treatment-related AEs were considered by the investigator to be possibly or probably related to study drug.
Time Frame: From date of first dose of study drug up to 30 days after the last dose of study drug, up to approximately 3 years
Population: Safety analysis set included all participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | 60 mg Placebo (Lower Baseline Platelet Count) | 60 mg Avatrombopag, (Lower Baseline Platelet Count) | 40 mg Placebo (Higher Baseline Platelet Count) | 40 mg Avatrombopag (Higher Baseline Platelet Count)
Number analyzed (Participants) | 48 | 89 | 32 | 58
Participants
  TEAEs | 31 | 53 | 18 | 31
  Treatment-related TEAEs | 7 | 12 | 2 | 4
  Serious TEAEs | 11 | 10 | 1 | 8
  TEAEs leading to study drug dose adjustment | 0 | 2 | 0 | 0
  TEAEs leading to study drug withdrawal | 0 | 2 | 0 | 0
  TEAEs leading to study drug dose reduction | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From date of administration of first dose up to 30 days after the last dose, up to approximately 3 years
Description: Treatment-emergent adverse events and all serious adverse events were reported. Adverse events were graded using Common Terminology Criteria for Adverse Event version 4. Safety analysis set included all participants who received at least 1 dose of study drug and had at least 1 post dose safety assessment. This set was analyzed "as treated".
Arm/Group | 60 mg Placebo (Lower Baseline Platelet Count) | 60 mg Avatrombopag, (Lower Baseline Platelet Count) | 40 mg Placebo (Higher Baseline Platelet Count) | 40 mg Avatrombopag (Higher Baseline Platelet Count)
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/89 | 0/32 | 2/58
Serious Adverse Events (participants affected / at risk) | 11/48 | 10/89 | 1/32 | 8/58
Other Adverse Events (participants affected / at risk) | 13/48 | 28/89 | 9/32 | 16/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 60 mg Placebo (Lower Baseline Platelet Count) (N=48) | 60 mg Avatrombopag, (Lower Baseline Platelet Count) (N=89) | 40 mg Placebo (Higher Baseline Platelet Count) (N=32) | 40 mg Avatrombopag (Higher Baseline Platelet Count) (N=58)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Splenomeglay (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Stress polycythaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0
Multiple Organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1
Chronic hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0
Clostridium test positive (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Coma hepatic (Nervous system disorders) | 0 | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 60 mg Placebo (Lower Baseline Platelet Count) (N=48) | 60 mg Avatrombopag, (Lower Baseline Platelet Count) (N=89) | 40 mg Placebo (Higher Baseline Platelet Count) (N=32) | 40 mg Avatrombopag (Higher Baseline Platelet Count) (N=58)
Abdominal pain (Gastrointestinal disorders) | 3 | 8 | 3 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 2 | 5
Fatigue (General disorders) | 1 | 6 | 1 | 1
Oedema peripheral (General disorders) | 2 | 3 | 1 | 3
Pyrexia (General disorders) | 5 | 7 | 1 | 5
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 6 | 0 | 0
Headache (Nervous system disorders) | 3 | 5 | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-12-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT01972529/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT01972529/SAP_001.pdf